CLINICAL TRIAL: NCT04064684
Title: Inhaled Steroids for the Treatment of Early Pediatric Acute Respiratory Distress Syndrome (PARDS), a Randomized Pilot Trial
Brief Title: Inhaled Steroids for the Treatment of Early Pediatric Acute Respiratory Distress Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment difficulties after the start of the COVID-19 pandemic.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Alvaro J Coronado Munoz, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-19-0566; KL2TR003168 (NIH)
Record Dates: First submitted 2019-08-16; First posted 2019-08-22 (Actual); Results first posted 2022-05-31 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-06

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Pediatric acute respiratory distress syndrome; PARDS; Budesonide; inhaled steroids
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Budesonide; Nebulizers and Vaporizers

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Budesonide administered by nebulizer (Experimental)
  Interventions: Drug: Budesonide; Device: Nebulizer
- Placebo administered by nebulizer (Placebo Comparator)
  Interventions: Drug: Placebo; Device: Nebulizer

INTERVENTIONS:
Drug: Budesonide — Enrolled patients will be treated with Pulmicort Respules® (Budesonide inhalation suspension), at a dose of 0.5 mg, nebulized twice daily through the mechanical ventilator. The medication will be administered to the patient by the respiratory therapist with the single-patient-use medication nebulizer attached to the mechanical ventilator circuit. The maximum length of treatment will be 10 days.
  Other Names: Pulmicort Respules®
  Arms: Budesonide administered by nebulizer
Drug: Placebo — Enrolled patients will be treated with normal saline.The medication will be administered to the patient by the respiratory therapist with the single-patient-use medication nebulizer attached to the mechanical ventilator circuit. The maximum length of treatment will be 10 days.
  Arms: Placebo administered by nebulizer
Device: Nebulizer — The medication will be administered to the patient by the respiratory therapist with the single-patient-use medication nebulizer attached to the mechanical ventilator circuit.

SUMMARY:
The purpose of this study is to show that inhaled steroids in patient with PARDS can decrease the days on mechanical ventilator measured by ventilator-free days,to improve the oxygenation index (OI) or oxygenation saturation index (OSI) in patients receiving inhaled steroids and to show the relevance and feasibility of a larger study by assessing the hypothesis in a small cohort of patients. Patient will be treated for a maximum of 10 days. Secondary objectives are to reduce the length of stay (LOS) in the pediatric intensive care unit (PICU) and hospital admissions; to show less inflammation in the patients receiving inhaled steroids by measuring inflammatory markers from tracheal aspirates like Interleukin (IL6, IL8, tumor necrosis factor (TNF) α, matrix metalloproteinase8 (MMP8) and matrix metalloproteinase9 (MMP9). Lastly, to show that inhaled steroids can improve residual lung disease evaluated by Pulmonary Function Test (PFTs) and Impulse Oscillometry (IOS).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients older than 30 days and up to 18 years of age admitted to the PICU with a diagnosis of PARDS enrolled within 72 hours of diagnosis.
* Patients requiring invasive mechanical ventilation.
* Criteria of PARDS as defined by the Pediatric Acute Lung Injury Consensus Conference (PALICC), on June 2015 in Pediatric Critical Care Journal

Exclusion Criteria:

* Patients with diffuse alveolar hemorrhage.
* Patients terminally ill with limitation of care or in hospice care.
* Patients receiving inhaled steroids or systemic steroids as chronic therapy before admission.
* Patients with high dose systemic steroids for anti-inflammatory purposes. The investigators will not exclude patients receiving hydrocortisone for shock.

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro J Coronado Munoz, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: months] | 6 (0) | 4 (0) | 5 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Ventilator-free Days (VFD)
Time Frame: Between the time of enrollment and day 28 after enrollment
Measure: Number; unit: days
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 1 | 1
days | 20 | 17

2. Secondary Outcome: Oxygenation Index (OI)
Description: Oxygenation index (OI) is calculated as ([FiO2 x Mean Airway Pressure] / PaO2). FiO2 stands for inspired fraction of oxygen, and PaO2 stands for pressure/arterial pressure of oxygen. An oxygenation index of 4-8 indicates mild ARDS, an oxygenation index of 8-16 indicates moderate ARDS, and an oxygenation index greater than 16 indicates severe ARDS.
Time Frame: Day one to last day of last day of mechanical ventilation (up to 10 days)
Population: For the participant in the budesonide arm, data for this outcome measure was not collected on days 9 and 10.
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 1 | 1
index
  day 1 | 11 (0) | 12 (0)
  day 2 | 11 (0) | 8 (0)
  day 3 | 8 (0) | 11.4 (0)
  day 4 | 4 (0) | 6.4 (0)
  day 5 | 3.2 (0) | 14.4 (0)
  day 6 | 3.5 (0) | 11.5 (0)
  day 7 | 5 (0) | 10 (0)
  day 8 | 2.8 (0) | 8.7 (0)
  day 9: number analyzed (Participants) | 0 | 1
  day 9 |  | 5 (0)
  day 10: number analyzed (Participants) | 0 | 1
  day 10 |  | 5 (0)

3. Secondary Outcome: Oxygen Saturation Index (OSI)
Description: 5-7.5 mild ARDS, 7.5-12.3 moderate ARDS. > 12.3 severe ARDS, formula FiO2*Mean airway pressure/Saturation of O2
  Oxygen saturation index (OI) is calculated as ([FiO2 x Mean Airway Pressure] / Saturation of oxygen). FiO2 stands for inspired fraction of oxygen. An oxygen saturation index of 5-7.5 indicates mild ARDS, an oxygen saturation index of 7.5-12.3 indicates moderate ARDS, and an oxygen saturation index greater than 12.3 indicates severe ARDS.
Time Frame: Day one to last day of last day of mechanical ventilation up to 28 days since enrollment
Population: Data for this outcome measure were not collected for either participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Days Participant Stayed in Pediatric Intensive Care Unit (PICU)
Time Frame: from time of enrollment until participant is transferred, discharged, or deceased (up to 50 days)
Measure: Number; unit: days
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 1 | 1
days | 46 | 17

5. Secondary Outcome: Number of Days Participant Stayed in Hospital
Time Frame: from time of enrollment until participant is transferred, discharged, or deceased (up to 50 days)
Measure: Number; unit: days
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 1 | 1
days | 46 | 23

6. Secondary Outcome: TNF Alpha Levels as Assessed by the Enzyme-linked Immunosorbent Assay (ELISA) Test
Time Frame: Day 1
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: TNF Alpha Levels as Assessed by the Enzyme-linked Immunosorbent Assay (ELISA) Test
Time Frame: Day 3
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: TNF Alpha Levels as Assessed by the Enzyme-linked Immunosorbent Assay (ELISA) Test
Time Frame: last day of treatment or last day of invasive mechanical ventilation( upto day 28)
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Interleukin (IL) -6 Levels as Assessed by the Enzyme-linked Immunosorbent Assay (ELISA) Test
Time Frame: Day 1
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: IL-6 Levels as Assessed by the Enzyme-linked Immunosorbent Assay (ELISA) Test
Time Frame: Day 3
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: IL-6 Levels as Assessed by the Enzyme-linked Immunosorbent Assay (ELISA) Test
Time Frame: last day of treatment or last day of invasive mechanical ventilation( upto day 28)
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: IL-8 Levels as Assessed by the Enzyme-linked Immunosorbent Assay (ELISA) Test
Time Frame: Day 1
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: IL-8 Levels as Assessed by the Enzyme-linked Immunosorbent Assay (ELISA) Test
Time Frame: Day 3
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: IL-8 Levels as Assessed by the Enzyme-linked Immunosorbent Assay (ELISA) Test
Time Frame: last day of treatment or last day of invasive mechanical ventilation( upto day 28)
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: MMP-8 Levels as Assessed by the Enzyme-linked Immunosorbent Assay (ELISA) Test
Time Frame: Day 1
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: MMP-8 Levels as Assessed by the Enzyme-linked Immunosorbent Assay (ELISA) Test
Time Frame: Day 3
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: MMP-8 Levels as Assessed by the Enzyme-linked Immunosorbent Assay (ELISA) Test
Time Frame: last day of treatment or last day of invasive mechanical ventilation( upto day 28)
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: MMP-9 Levels as Assessed by the Enzyme-linked Immunosorbent Assay (ELISA) Test
Time Frame: Day 1
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: MMP-9 Levels as Assessed by the Enzyme-linked Immunosorbent Assay (ELISA) Test
Time Frame: Day 3
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: MMP-9 Levels as Assessed by the Enzyme-linked Immunosorbent Assay (ELISA) Test
Time Frame: last day of treatment or last day of invasive mechanical ventilation( upto day 28)
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Neutrophil Count
Time Frame: Day 1
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Neutrophil Count
Time Frame: Day 3
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Neutrophil Count
Time Frame: last day of treatment or last day of invasive mechanical ventilation( upto day 28)
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: FEV1
Description: Forced expiration in 1st second, abnormal (obstructive)<80% L/second
Time Frame: 90 days since first day of treatment
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Forced Expiratory Volume at One Second FEV1/FVC
Description: Restrictive disease if <70%
Time Frame: 90 days since first day of treatment
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Forced Vital Capacity (FVC)
Description: <80% restrictive lung disease, L
Time Frame: 90 days since first day of treatment
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Forced Expiratory Flow FEF 25-75%
Description: Medium size bronchioles, normal 60-130%
Time Frame: 90 days since first day of treatment
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Respiratory Resistance by Impulse Oscillometry (IOS)
Description: Rrs 3-35 Hz
Time Frame: 90 days since first day of treatment
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Respiratory Impedance by Impulse Oscillometry (IOS)
Description: Zrs 3-35 Hz
Time Frame: 90 days since first day of treatment
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Respiratory Reactance by Impulse Oscillometry (IOS)
Description: Xrs 3-35 Hz
Time Frame: 90 days since first day of treatment
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Budesonide Administered by Nebulizer | Placebo Administered by Nebulizer
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Enrollment difficulties after start of the COVID-19 pandemic leading to small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT04064684/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT04064684/ICF_001.pdf